CLINICAL TRIAL: NCT06632184
Title: Pilot Comparative Study on the Efficacy of Multimodal Management With Peritoneal Lavage Using Saline Solution Versus Saline Solution With Ondansetron in Laparoscopic Cholecystectomy
Brief Title: Peritoneal Lavage Using Saline or Saline With Ondansetron for Pain Control After Laparoscopic Cholecystectomy
Acronym: PLUSO
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Francisco Aguilar Espinosa, General Surgery department: Dr. Francisco Aguilar Espinosa, Clinical Research, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F-CNIC-2024-097; R-2025-785-080 (Other: Instituto Mexicano del Seguro Social (IMSS))
Record Dates: First submitted 2024-10-05; First posted 2024-10-08 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Pain Management; Laparoscopic Cholecystectomy; Ondansetron; Postoperative Nausea and Vomiting
Keywords: Laparoscopic cholecystectomy; Ondansetron Formulations; Intraperitoneal Analgesia; Saline Solution; Pain Management; Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Agnosia | interventions — Ondansetron; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: nterventional Study Model: Parallel assignment. Participants are randomized into one of two parallel groups in a 1:1 ratio to receive either the experimental intervention or the control intervention for the duration of the study. The model incorporates triple-blinding (participant, care provider, outcomes assessor) and a randomized, controlled design. Allocation is performed using a computer-generated sequence with permuted blocks, stratified by sex and ASA physical status classification to ensure balanced groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a triple-blind study. Beyond the participant, the following key parties are masked: the surgeons performing the procedure, the anesthesiologists managing perioperative care, and the post-operative outcome assessors (e.g., research interns collecting pain scores and other clinical data). A designated "blinding coordination nurse," who is not involved in any clinical or assessment roles, prepares the identical-looking solutions according to the randomization sequence. The data analyst will also remain masked to group allocation (coded as A/B) until the completion of the primary statistical analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Saline Lavage Only (Active Comparator): Participants in this arm will receive intraoperative peritoneal lavage with 500 mL of 0.9% saline solution for 5 minutes at the end of laparoscopic cholecystectomy. The solution will be fully aspirated before abdominal closure. The solution will remain in the peritoneal cavity for 5 minutes and then be completely aspirated before closure. All participants will also receive standard multimodal analgesia including paracetamol, diclofenac, and local wound infiltration with bupivacaine.
  Interventions: Drug: Saline Intraperitoneal Lavage
- Saline Lavage With Ondansetron (Experimental): Participants in this arm will undergo peritoneal lavage with 500 mL of 0.9% saline solution combined with 8 mg of ondansetron, administered intraperitoneally at the end of elective laparoscopic cholecystectomy. The solution will remain in the peritoneal cavity for 5 minutes and then be completely aspirated before closure. All participants will also receive standard multimodal analgesia including paracetamol, diclofenac, and local wound infiltration with bupivacaine.
  Interventions: Drug: Ondansetron Intraperitoneal Lavage

INTERVENTIONS:
Drug: Ondansetron Intraperitoneal Lavage — A single dose of 8 mg of ondansetron diluted in 500 mL of 0.9% saline solution will be administered as an intraperitoneal lavage at the end of elective laparoscopic cholecystectomy. The solution will remain in the abdominal cavity for 5 minutes and then be fully aspirated before surgical closure. This intervention aims to evaluate the local analgesic and antiemetic effects of ondansetron when used via the peritoneal route.
  Other Names: Ondansetron; Zofran; 0.9% Sodium Chloride
  Arms: Saline Lavage With Ondansetron
Drug: Saline Intraperitoneal Lavage — At the end of elective laparoscopic cholecystectomy, a peritoneal lavage will be performed using 500 mL of 0.9% saline solution (normal saline). The solution will be maintained in the peritoneal cavity for 5 minutes and then fully aspirated before surgical closure. This intervention serves as the comparator to assess the added effect of ondansetron in the experimental group.
  Other Names: normal saline; 0.9% Sodium Chloride; Saline Solution
  Arms: Saline Lavage Only

SUMMARY:
Brief Summary Background: Laparoscopic cholecystectomy is a common procedure where postoperative pain and nausea/vomiting (PONV) remain significant issues, impairing recovery. Standardized multimodal analgesia (e.g., PROSPECT guidelines) is effective for pain, but PONV incidence stays high. Preliminary evidence suggests that adding ondansetron to the standard intraperitoneal saline lavage could provide additional analgesic and antiemetic benefits by blocking peripheral 5-HT3 receptors at the trauma site.

Objective: This pilot study aims to evaluate if intraperitoneal lavage with saline + 8mg ondansetron reduces the total burden of postoperative pain over the first 24 hours (Area Under the Curve of the Visual Analog Scale, AUC-VAS/24h) compared to saline lavage alone, within a standardized multimodal protocol.

Methods: This is a phase IV, pilot, randomized, controlled, triple-blind clinical trial. 40 adult patients (ASA I-II) undergoing elective laparoscopic cholecystectomy for symptomatic cholelithiasis (Nassar Grade I-II difficulty) will be randomly assigned (1:1) to:

Control Group: 500 ml of 0.9% saline intraperitoneal lavage.

Intervention Group: 500 ml of 0.9% saline + 8 mg ondansetron intraperitoneal lavage.

The lavage is performed for 5 minutes at the end of surgery, followed by complete aspiration. All patients receive a strict multimodal perioperative protocol, including pre-incisional port site infiltration with bupivacaine 0.75%, standardized anesthesia, and postoperative analgesics. The use of intravenous ondansetron is prohibited to avoid confounding.

Primary Outcome: Total postoperative pain burden (AUC-VAS/24h). Secondary Outcomes (Exploratory): PONV incidence; time to first rescue analgesia; rescue analgesic consumption (buprenorphine); postoperative sleep quality (Richards-Campbell Sleep Questionnaire); safety and adverse events.

DETAILED DESCRIPTION:
1. Study Rationale and Background Postoperative pain and PONV are prevalent after laparoscopic cholecystectomy, leading to patient discomfort, prolonged hospitalization, and increased resource use. The PROSPECT guidelines recommend a multimodal approach, including intraperitoneal saline lavage, to mitigate pain by diluting irritants and reducing acidosis. However, even with this approach, PONV rates remain high (30-50%).

   Ondansetron, a 5-HT3 antagonist, is a established antiemetic. Emerging evidence indicates a peripheral analgesic mechanism via blocking 5-HT3 receptors on nociceptive neurons, inhibiting neuropeptide release, and potential local anesthetic effects. Administering it intraperitoneally targets the site of surgical trauma. A previous study (Abdelaziz et al., 2021) using 4mg showed promise, but it had a small sample size and was not integrated into a strict, modern multimodal protocol. This pilot study addresses this gap by testing an 8mg dose within a rigorous, standardized PROSPECT-aligned protocol, using the AUC-VAS/24h to comprehensively capture the pain burden.
2. Overall Study Design and Methodology This is a single-center, prospective, phase IV, randomized, controlled, triple-blind, parallel-group pilot study, designed and reported according to CONSORT guidelines for pilot trials.

   Blinding (Triple):

   Patients are unaware of their assignment.

   Care Providers & Outcome Assessors: Surgeons, anesthesiologists, nurses, and research interns collecting data are all blinded.

   Data Analyst: The statistician performs the initial analysis on coded data (Group A/B) before unblinding.

   Randomization: A computer-generated sequence using permuted blocks (sizes 4 and 6), stratified by sex and ASA status (I vs. II), will allocate patients 1:1. Allocation is concealed using sequentially numbered, opaque, sealed envelopes. A designated "blinding coordination nurse" opens the envelope, prepares the identical-looking study solution, and labels it only with a code (A or B).
3. Standardization of Procedures A strict, standardized perioperative protocol is mandated for all participants to minimize variability.

   Preoperative:

   Dexamethasone 8mg IV (antiemetic), antibiotic prophylaxis.

   Intraoperative:

   Anesthesia: Standardized induction (Midazolam 0.02-0.03 mg/kg, Fentanyl 2-4 mcg/kg, Propofol 1-2 mg/kg, Cisatracurium 0.15 mg/kg) and maintenance (Sevoflurano 1-1.5 MAC). Multimodal analgesia: Acetaminophen 1g IV and Diclofenac 75mg IV.

   Surgery: Pneumoperitoneum pressure strictly maintained at 10-12 mmHg. Four-port technique with identical placement. Pre-incisional infiltration of all port sites with Bupivacaine 0.75% (up to 20 ml total). Critical view of safety dissection. Active and complete aspiration of pneumoperitoneum at closure.

   Intervention: The assigned solution (500ml) is instilled into the peritoneal cavity for 5 minutes with the patient in a 20° Trendelenburg position, followed by complete aspiration.

   Postoperative:

   Scheduled analgesics: Acetaminophen 1g (every 8 hours) and Diclofenac 75mg IV (every 12 hours).

   Rescue Analgesia: Buprenorphine 75mcg SC is administered only upon patient request AND a pain score ≥50mm on the VAS or ≥6 on the Faces Pain Scale-Revised (FPS-R).

   Rescue Antiemesis: Metoclopramida 10mg IV is permitted for PONV. The use of intravenous ondansetron is prohibited during the entire perioperative period to avoid confounding the intervention's effects.
4. Objectives and Endpoints as a Pilot Study As a pilot trial, its primary goal is to assess feasibility, refine procedures, and obtain preliminary estimates of effect and variability to power a future definitive trial. The primary outcome, AUC-VAS/24h, integrates pain intensity and duration, providing a robust measure of the "total pain burden." All secondary outcomes (PONV, rescue analgesia consumption, sleep quality) are explicitly exploratory and hypothesis-generating.
5. Safety and Monitoring The safety of intraperitoneal saline lavage and ondansetron is well-established. The combination presents minimal anticipated risk. All adverse events and postoperative complications will be actively monitored and recorded for the first 24 hours and up to 30 days post-surgery. An interim analysis for safety and efficacy will be conducted after 50% recruitment (n=20). Any serious adverse events will be reported promptly to the Institutional Ethics Committee.
6. Significance This is the first study to evaluate the combination of standard saline lavage with 8mg of intraperitoneal ondansetron within a rigorously standardized, PROSPECT-aligned, multimodal protocol. Using a triple-blind pilot design and a comprehensive primary endpoint, it will generate high-quality preliminary evidence on this simple, low-cost intervention's efficacy and safety in a Mexican population. The results will determine the feasibility and inform the design of a larger, definitive multicenter randomized controlled trial.

ELIGIBILITY:
Eligible participants will be adult patients scheduled for elective laparoscopic cholecystectomy at the study site. To ensure a homogeneous sample appropriate for this pilot trial, strict inclusion and exclusion criteria have been defined.

Inclusion criteria

Patients meeting all the following criteria will be considered for enrollment:

1. Aged between 18 and 60 years.
2. American Society of Anesthesiologist (ASA) physical status classification I or II.
3. Scheduled for elective laparoscopic cholecystectomy due to symptomatic cholelithiasis, resolved choledocholithiasis post-endoscopic retrograde cholangiopancreatography (ERCP), or gallbladder polyp.
4. Placement of a ¾-inch Penrose drain in the subhepatic cavity as part of the standardized surgical technique, to allow evacuation of residual CO2, residual lavage fluid, and close monitoring for possible postoperative bleeding or bile leakage.
5. Intraoperative surgical difficulty assessed as Grade I, II or III according to the Nassar scale
6. Ability to provide written, informed consent

Exclusion Criteria

Patients presenting with any of the following will be excluded:

1. Confirmed pregnancy or lactation
2. Intraoperative findings of Nassar Grade IV, suspected gallbladder cancer, scleroatrophic gallbladder, or cirrhosis

5. Use of NSAIDs within 24 hours prior to surgery, or chronic use of NSAIDs, opioids, immunosuppressants, chemotherapy, or anticoagulants.

6. Known allergies to ondansetron, acetaminophen, diclofenac sodium, buprenorphine or tramadol

7. Significant cardiac disease (e.g., heart failure, arrhythmias, pacemaker dependency)

8. Obesity Grade IV (Body Mass Index ≥ 50 kg/m2)

9. History of recurrent vertigo or motion sickness

Elimination Criteria

Patients who meet inclusion criteria but experience the following intraoperative events will be eliminated from the final per-protocol analysis: significant bleeding or bile duct injury requiring re-intervention, conversion to open surgery, or a total operative time exceeding 80 minutes.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Total Pain Burden as Measured by the Area Under the Curve (AUC) of Visual Analog Scale (VAS) Scores Over the First 24 Postoperative Hours | 0, 2, 6, 12, and 24 hours postoperatively
  The primary outcome is the total burden of postoperative pain, quantified as the Area Under the Curve (AUC) of serial Visual Analog Scale (VAS) scores measured at 0, 2, 6, 12, and 24 hours after surgery. The AUC is calculated using the trapezoidal rule, which integrates both the intensity and duration of pain into a single composite measure (units: mm*hour). This provides a more comprehensive assessment of the patient's pain experience over the critical first postoperative day than isolated time-point measurements. A lower AUC indicates superior pain control.

SECONDARY OUTCOMES:
Incidence of Postoperative Nausea and Vomiting (PONV) | 0, 2, 6, 12, and 24 hours postoperatively
  The presence and number of postoperative nausea and vomiting (PONV)
Use of Rescue Analgesia Within 24 Hours Postoperatively | 0 to 24 hours postoperatively
  The proportion of patients requiring rescue analgesia (buprenorphine 75 mcg subcutaneously) will be recorded. The time to first dose and the total number of doses will also be analyzed.
Postoperative Sleep Quality Assessed by the Richards-Campbell Sleep Questionnaire | Night of surgery to morning after surgery
  Sleep quality will be evaluated using the Richards-Campbell Sleep Questionnaire, which includes six visual analog items rated from 0 to 100. A higher score indicates better sleep. The total average score will be calculated for each participant.
Incidence of Adverse Events Possibly Related to Intraperitoneal Ondansetron | 0 to 24 hours postoperatively
  Any unexpected clinical signs, symptoms, or laboratory abnormalities that could be associated with the intraperitoneal use of ondansetron will be recorded and evaluated by the study team.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Aguilar Espinosa, Dr., Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- General Hospital No. 89 of the Mexican Social Security Institute (IMSS), Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share individual participant data (IPD) has not yet been finalized. Data sharing will depend on the outcomes of the pilot study, ethical considerations, and institutional policies. Any future data sharing will ensure patient confidentiality and comply with regulatory standards.

REFERENCES:
- [Result] Subhas G, Gupta A, Bhullar J, Dubay L, Ferguson L, Goriel Y, Jacobs MJ, Kolachalam RB, Silapaswan S, Mittal VK. Prolonged (longer than 3 hours) laparoscopic cholecystectomy: reasons and results. Am Surg. 2011 Aug;77(8):981-4. PMID 21944510
- [Result] Wang DE, Bakshi C, Sugiyama G, Coppa G, Alfonso A, Chung P. Does Operative Time Affect Complication Rate in Laparoscopic Cholecystectomy. Am Surg. 2023 Nov;89(11):4479-4484. doi: 10.1177/00031348221117032. Epub 2022 Aug 11. PMID 38050322
- [Result] Rudasill SE, Dillon D, Karunungan K, Mardock AL, Hadaya J, Sanaiha Y, Tran Z, Benharash P. The obesity paradox: Underweight patients are at the greatest risk of mortality after cholecystectomy. Surgery. 2021 Sep;170(3):675-681. doi: 10.1016/j.surg.2021.03.034. Epub 2021 Apr 28. PMID 33933284
- [Result] Reeves JJ, Burton BN, Broderick RC, Waterman RS, Gabriel RA. Obesity and unanticipated hospital admission following outpatient laparoscopic cholecystectomy. Surg Endosc. 2021 Mar;35(3):1348-1354. doi: 10.1007/s00464-020-07514-7. Epub 2020 Mar 23. PMID 32206919
- [Result] Augustin T, Moslim MA, Brethauer S, Aminian A, Kroh M, Schneider E, Walsh RM. Obesity and its implications for morbidity and mortality after cholecystectomy: A matched NSQIP analysis. Am J Surg. 2017 Mar;213(3):539-543. doi: 10.1016/j.amjsurg.2016.11.037. Epub 2017 Jan 26. PMID 28237044
- [Result] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Result] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Result] Miranda-Ackerman RC, Lira-Trujillo M, Gollaz-Cervantez AC, Cortes-Flores AO, Zuloaga-Fernandez Del Valle CJ, Garcia-Gonzalez LA, Morgan-Villela G, Barbosa-Camacho FJ, Pintor-Belmontes KJ, Guzman-Ramirez BG, Bernal-Hernandez A, Fuentes-Orozco C, Gonzalez-Ojeda A. Associations between stressors and difficulty sleeping in critically ill patients admitted to the intensive care unit: a cohort study. BMC Health Serv Res. 2020 Jul 9;20(1):631. doi: 10.1186/s12913-020-05497-8. PMID 32646516
- [Result] Garcia-Galicia A, Guzman-Maya I, Montiel-Jarquin AJ, Parra-Salazar JA, Gonzalez-Lopez AM, Loria-Castellanos J. Validation of a faces pain scale in postsurgical geriatric patients. Cir Cir. 2021;89(2):212-217. doi: 10.24875/CIRU.20000094. PMID 33784276
- [Result] Sandoval-Jimenez CH, Mendez-Sashida GJ, Cruz-Marquez-Rico LM, Cardenas-Victorica R, Guzman-Esquivel H, Luna-Silva M, Diaz-Valero R. [Postoperative pain in patients undergoing elective laparoscopic cholecystectomy with low versus standard-pressure pneumoperitoneum. A randomized clinical trial.]. Rev Gastroenterol Mex. 2009 Oct-Dec;74(4):314-20. Spanish. PMID 20423760
- [Result] Reddi BA. Why is saline so acidic (and does it really matter?). Int J Med Sci. 2013 Apr 17;10(6):747-50. doi: 10.7150/ijms.5868. Print 2013. PMID 23630439
- [Result] Graham CL, Dukes GE, Kao CF, Bertch JM, Hak LJ. Stability of ondansetron in large-volume parenteral solutions. Ann Pharmacother. 1992 Jun;26(6):768-71. doi: 10.1177/106002809202600603. PMID 1535245
- [Result] Zhang D, Wang X, Yang X, Xia D. The effect of intraperitoneal instillation of drugs on postoperative analgesia after laparoscopic cholecystectomy: a network meta-analysis. Front Pharmacol. 2025 Sep 12;16:1646917. doi: 10.3389/fphar.2025.1646917. eCollection 2025. PMID 41020002
- [Result] Sravanthi GC, Abuji K, Soni SL, Nagaraj SS, Sharma A, Jafra A, Tandup C, Kurdia KC, Dahiya D. Effect of intraperitoneal magnesium sulfate in the prevention of postoperative pain in daycare laparoscopic cholecystectomy - A prospective randomized controlled trial. Indian J Pharmacol. 2023 May-Jun;55(3):174-178. doi: 10.4103/ijp.ijp_827_22. PMID 37555412
- [Result] Vijayaraghavalu S, Bharthi Sekar E. A Comparative Study on the Postoperative Analgesic Effects of the Intraperitoneal Instillation of Bupivacaine Versus Normal Saline Following Laparoscopic Cholecystectomy. Cureus. 2021 Mar 27;13(3):e14151. doi: 10.7759/cureus.14151. PMID 33927953
- [Result] Rahimzadeh P, Faiz SHR, Hoseini M, Mousavie SH, Imani F, Negah AR. Comparison of intraperitoneal bupivacaine, acetazolamide, and placebo on pain relief after laparoscopic cholecystectomy surgery: A clinical trial. Med J Islam Repub Iran. 2018 Nov 13;32:112. doi: 10.14196/mjiri.32.112. eCollection 2018. PMID 30815407
- [Result] Putta PG, Pasupuleti H, Samantaray A, Natham H, Rao MH. A comparative evaluation of pre-emptive versus post-surgery intraperitoneal local anaesthetic instillation for postoperative pain relief after laparoscopic cholecystectomy: A prospective, randomised, double blind and placebo controlled study. Indian J Anaesth. 2019 Mar;63(3):205-211. doi: 10.4103/ija.IJA_767_18. PMID 30988535
- [Result] Nikoubakht N, Faiz SHR, Mousavie SH, Shafeinia A, Borhani Zonoz L. Effect of bupivacaine intraperitoneal and intra-abdominal bicarbonate in reducing postoperative pain in laparoscopic cholecystectomy: a double-blind randomized clinical trial study. BMC Res Notes. 2022 Jun 3;15(1):191. doi: 10.1186/s13104-022-06083-3. PMID 35659713
- [Result] Melidi E, Papadima A, Pandazi A, Zografos G. Efficacy of Repeated Intraperitoneal Administration of Levobupivacaine in Pain and Opioid Consumption After Elective Laparoscopic Cholecystectomy: A Prospective Randomized Placebo-controlled Trial. Surg Laparosc Endosc Percutan Tech. 2016 Aug;26(4):295-300. doi: 10.1097/SLE.0000000000000297. PMID 27380615
- [Result] Honca M, Kose EA, Bulus H, Horasanli E. The postoperative analgesic efficacy of intraperitoneal bupivacaine compared with levobupivacaine in laparoscopic cholecystectomy. Acta Chir Belg. 2014 May-Jun;114(3):174-8. doi: 10.1080/00015458.2014.11681004. PMID 25102706
- [Result] Labaille T, Mazoit JX, Paqueron X, Franco D, Benhamou D. The clinical efficacy and pharmacokinetics of intraperitoneal ropivacaine for laparoscopic cholecystectomy. Anesth Analg. 2002 Jan;94(1):100-5, table of contents. doi: 10.1097/00000539-200201000-00019. PMID 11772809
- [Result] Abdelhedi A, Ketata S, Kardoun N, Keskes M, Zouche I, Ayedi A, Doukeli O, Khrouf M, Fendri S, Zouari A, Cheikhrouhou H. [The effect of intraperitoneal administration of dexamethasone on postoperative analgesia after laparoscopic cholecystectomy: a prospective randomized controlled double-blind study]. Pan Afr Med J. 2023 May 4;45:14. doi: 10.11604/pamj.2023.45.14.36438. eCollection 2023. French. PMID 37426459
- [Result] Kaushal-Deep SM, Anees A, Khan S, Khan MA, Lodhi M. Randomized controlled study of intraincisional infiltration versus intraperitoneal instillation of standardized dose of ropivacaine 0.2% in post-laparoscopic cholecystectomy pain: Do we really need high doses of local anesthetics-time to rethink! Surg Endosc. 2018 Jul;32(7):3321-3341. doi: 10.1007/s00464-018-6053-z. Epub 2018 Jan 16. PMID 29340809
- [Result] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Result] Al Shoyaib A, Archie SR, Karamyan VT. Intraperitoneal Route of Drug Administration: Should it Be Used in Experimental Animal Studies? Pharm Res. 2019 Dec 23;37(1):12. doi: 10.1007/s11095-019-2745-x. PMID 31873819
- [Result] Roila F, Del Favero A. Ondansetron clinical pharmacokinetics. Clin Pharmacokinet. 1995 Aug;29(2):95-109. doi: 10.2165/00003088-199529020-00004. PMID 7586904
- [Result] Skovgard K, Agerskov C, Kohlmeier KA, Herrik KF. The 5-HT3 receptor antagonist ondansetron potentiates the effects of the acetylcholinesterase inhibitor donepezil on neuronal network oscillations in the rat dorsal hippocampus. Neuropharmacology. 2018 Dec;143:130-142. doi: 10.1016/j.neuropharm.2018.09.017. Epub 2018 Sep 19. PMID 30243914
- [Result] McCleane GJ, Suzuki R, Dickenson AH. Does a single intravenous injection of the 5HT3 receptor antagonist ondansetron have an analgesic effect in neuropathic pain? A double-blinded, placebo-controlled cross-over study. Anesth Analg. 2003 Nov;97(5):1474-1478. doi: 10.1213/01.ANE.0000085640.69855.51. PMID 14570668
- [Result] Li CJ, Zhang LG, Liu LB, An MQ, Dong LG, Gu HY, Dai YP, Wang F, Mao CJ, Liu CF. Inhibition of Spinal 5-HT3 Receptor and Spinal Dorsal Horn Neuronal Excitability Alleviates Hyperalgesia in a Rat Model of Parkinson's Disease. Mol Neurobiol. 2022 Dec;59(12):7253-7264. doi: 10.1007/s12035-022-03034-8. Epub 2022 Sep 27. PMID 36168076
- [Result] Khasabov SG, Lopez-Garcia JA, Asghar AU, King AE. Modulation of afferent-evoked neurotransmission by 5-HT3 receptors in young rat dorsal horn neurones in vitro: a putative mechanism of 5-HT3 induced anti-nociception. Br J Pharmacol. 1999 Jun;127(4):843-52. doi: 10.1038/sj.bjp.0702592. PMID 10433490
- [Result] Ye JH, Mui WC, Ren J, Hunt TE, Wu WH, Zbuzek VK. Ondansetron exhibits the properties of a local anesthetic. Anesth Analg. 1997 Nov;85(5):1116-21. doi: 10.1097/00000539-199711000-00029. PMID 9356111
- [Result] Khoori M, Mirghaderi P, Azarboo A, Jamil F, Eshraghi N, Baghaei AA. Effect of Ondansetron on Postoperative Pain and Vomiting after Acute Appendicitis Surgery: A Placebo-Controlled Double-Blinded Randomized Clinical Trial. Pain Res Manag. 2024 Jun 12;2024:6429874. doi: 10.1155/2024/6429874. eCollection 2024. PMID 38899063
- [Result] Ye JH, Ponnudurai R, Schaefer R. Ondansetron: a selective 5-HT(3) receptor antagonist and its applications in CNS-related disorders. CNS Drug Rev. 2001 Summer;7(2):199-213. doi: 10.1111/j.1527-3458.2001.tb00195.x. PMID 11474424
- [Result] Giordano J, Dyche J. Differential analgesic actions of serotonin 5-HT3 receptor antagonists in the mouse. Neuropharmacology. 1989 Apr;28(4):423-7. doi: 10.1016/0028-3908(89)90040-3. PMID 2526302
- [Result] Zeitz KP, Guy N, Malmberg AB, Dirajlal S, Martin WJ, Sun L, Bonhaus DW, Stucky CL, Julius D, Basbaum AI. The 5-HT3 subtype of serotonin receptor contributes to nociceptive processing via a novel subset of myelinated and unmyelinated nociceptors. J Neurosci. 2002 Feb 1;22(3):1010-9. doi: 10.1523/JNEUROSCI.22-03-01010.2002. PMID 11826129
- [Result] Sufka KJ, Schomburg FM, Giordano J. Receptor mediation of 5-HT-induced inflammation and nociception in rats. Pharmacol Biochem Behav. 1992 Jan;41(1):53-6. doi: 10.1016/0091-3057(92)90058-n. PMID 1531705
- [Result] Farouk S. Ondansetron added to lidocaine for intravenous regional anaesthesia. Eur J Anaesthesiol. 2009 Dec;26(12):1032-6. doi: 10.1097/EJA.0b013e3283317d93. PMID 19707145
- [Result] Wolf H. Preclinical and clinical pharmacology of the 5-HT3 receptor antagonists. Scand J Rheumatol Suppl. 2000;113:37-45. doi: 10.1080/030097400446625. PMID 11028830
- [Result] Rusch D, Eberhart LH, Wallenborn J, Kranke P. Nausea and vomiting after surgery under general anesthesia: an evidence-based review concerning risk assessment, prevention, and treatment. Dtsch Arztebl Int. 2010 Oct;107(42):733-41. doi: 10.3238/arztebl.2010.0733. Epub 2010 Oct 22. PMID 21079721
- [Result] Gan TJ. Risk factors for postoperative nausea and vomiting. Anesth Analg. 2006 Jun;102(6):1884-98. doi: 10.1213/01.ANE.0000219597.16143.4D. PMID 16717343
- [Result] Wills VL, Hunt DR. Pain after laparoscopic cholecystectomy. Br J Surg. 2000 Mar;87(3):273-84. doi: 10.1046/j.1365-2168.2000.01374.x. PMID 10718794
- [Result] Mouton WG, Bessell JR, Otten KT, Maddern GJ. Pain after laparoscopy. Surg Endosc. 1999 May;13(5):445-8. doi: 10.1007/s004649901011. PMID 10227938
- [Result] Bisgaard T, Kehlet H, Rosenberg J. Pain and convalescence after laparoscopic cholecystectomy. Eur J Surg. 2001 Feb;167(2):84-96. doi: 10.1080/110241501750070510. PMID 11266262
- [Result] Barazanchi AWH, MacFater WS, Rahiri JL, Tutone S, Hill AG, Joshi GP; PROSPECT collaboration. Evidence-based management of pain after laparoscopic cholecystectomy: a PROSPECT review update. Br J Anaesth. 2018 Oct;121(4):787-803. doi: 10.1016/j.bja.2018.06.023. Epub 2018 Aug 7. PMID 30236241
- [Result] Abdelaziz DH, Boraii S, Cheema E, Elnaem MH, Omar T, Abdelraouf A, Mansour NO. The intraperitoneal ondansetron for postoperative pain management following laparoscopic cholecystectomy: A proof-of-concept, double-blind, placebo-controlled trial. Biomed Pharmacother. 2021 Aug;140:111725. doi: 10.1016/j.biopha.2021.111725. Epub 2021 May 18. PMID 34015580
- [Result] Ko-Iam W, Paiboonworachat S, Pongchairerks P, Junrungsee S, Sandhu T. Combination of etoricoxib and low-pressure pneumoperitoneum versus standard treatment for the management of pain after laparoscopic cholecystectomy: a randomized controlled trial. Surg Endosc. 2016 Nov;30(11):4800-4808. doi: 10.1007/s00464-016-4810-4. Epub 2016 Feb 23. PMID 26905574
- [Result] Kim HC, Song Y, Lee JS, Jeong ME, Lee Y, Lim JH, Kim DH. Comparison of pharmacologic therapies alone versus operative techniques in combination with pharmacologic therapies for postoperative analgesia in patients undergoing laparoscopic cholecystectomy: A randomized controlled trial. Int J Surg. 2022 Aug;104:106763. doi: 10.1016/j.ijsu.2022.106763. Epub 2022 Jul 6. PMID 35803512
- [Result] Seo YK, Lee HJ, Ha TK, Lee KG. Effect of normal saline irrigation on attenuation of shoulder tip pain and on beta-endorphin levels after laparoscopic cholecystectomy. J Laparoendosc Adv Surg Tech A. 2012 May;22(4):311-4. doi: 10.1089/lap.2011.0365. Epub 2012 Jan 30. PMID 22288883
- [Result] Bala I, Bhatia N, Mishra P, Verma GR, Kaman L. Comparison of preoperative oral acetazolamide and intraperitoneal normal saline irrigation for reduction of postoperative pain after laparoscopic cholecystectomy. J Laparoendosc Adv Surg Tech A. 2015 Apr;25(4):285-90. doi: 10.1089/lap.2014.0507. Epub 2015 Mar 13. PMID 25768238
- [Result] Barthelsson C, Sandblom G, Ljesevic-Nikoletic S, Hammarqvist F. Effects of Intra-abdominally Instilled Isotonic Saline on Pain, Recovery, and Health-Related Quality-of-Life Following Laparoscopic Cholecystectomy: A Randomized Prospective Double-Blind Controlled Study. World J Surg. 2015 Jun;39(6):1413-20. doi: 10.1007/s00268-015-2978-8. PMID 25665674
- [Result] Allen RW, Burney CP, Davis A, Henkin J, Kelly J, Judd BG, Ivatury SJ. Deep Sleep and Beeps: Sleep Quality Improvement Project in General Surgery Patients. J Am Coll Surg. 2021 Jun;232(6):882-888. doi: 10.1016/j.jamcollsurg.2021.02.010. Epub 2021 Mar 3. PMID 33675989
- [Result] Abdelraheem Mohamed M, Elsayed HM, Badawy FA. A comparative study of the analgesic efficacy of intraperitoneal instillation of diluted bupivacaine versus non-diluted bupivacaine after laparoscopic cholecystectomy: a prospective single-blinded controlled randomized study. Egypt J Anaesth. 2023;39(1):1-6.
- [Result] Awolaran O, Gana T, Samuel N, Oaikhinan K. Readmissions after laparoscopic cholecystectomy in a UK District General Hospital. Surg Endosc. 2017 Sep;31(9):3534-3538. doi: 10.1007/s00464-016-5380-1. Epub 2016 Dec 23. PMID 28008467
- [Result] Moghadamyeghaneh Z, Badami A, Masi A, Misawa R, Dresner L. Unplanned readmission after outpatient laparoscopic cholecystectomy. HPB (Oxford). 2020 May;22(5):702-709. doi: 10.1016/j.hpb.2019.09.005. Epub 2019 Sep 28. PMID 31575471
- [Result] Rosero EB, Joshi GP. Hospital readmission after ambulatory laparoscopic cholecystectomy: incidence and predictors. J Surg Res. 2017 Nov;219:108-115. doi: 10.1016/j.jss.2017.05.071. Epub 2017 Jun 28. PMID 29078868
- [Result] Keus F, de Jong JA, Gooszen HG, van Laarhoven CJ. Laparoscopic versus small-incision cholecystectomy for patients with symptomatic cholecystolithiasis. Cochrane Database Syst Rev. 2006 Oct 18;2006(4):CD006229. doi: 10.1002/14651858.CD006229. PMID 17054284
- [Result] Mendez Sanchez N, Uribe Esquivel M, Jessurun Solomou J, Cervera Ceballos E, Bosques Padilla F. [Epidemiology of gallstone disease in Mexico]. Rev Invest Clin. 1990 Jul;42 Suppl:48-52. Spanish. PMID 19256134
- [Result] Cobos-Carbo A; CONSORT group. [Randomized clinical trials (CONSORT)]. Med Clin (Barc). 2005 Dec 1;125 Suppl 1:21-7. doi: 10.1016/s0025-7753(05)72205-3. Spanish. PMID 16464423

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-11-13): https://cdn.clinicaltrials.gov/large-docs/84/NCT06632184/Prot_SAP_ICF_001.pdf